CLINICAL TRIAL: NCT05179395
Title: Brasthesis Prototype for Women Veterans With Upper Limb Amputations
Brief Title: Brasthesis Prosthetic Harness for Women Veterans With Upper Limb Amputations
Acronym: Brasthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: A3851-P; I21RX003851-01A1 (NIH)
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Upper Limb Amputation
Keywords: amputation; artificial limb

STUDY DESIGN:
Intervention Model Description: All Participants unilateral upper limb amputation participants will wear the Brasthesis harness with their prosthetic arm for 4 weeks. Each subject served as their own control with baseline data collected at visit 1 and interventional data collected after 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Brasthesis (Experimental): All five participants will wear Brasthesis for 4-weeks
  Interventions: Device: Brasthesis

INTERVENTIONS:
Device: Brasthesis — Brasthesis is a harness that is integrated with an off the shelf sports bra

SUMMARY:
This project tests Brasthesis, a new product for women Veterans with upper limb loss. Brasthesis incorporates the harnessing straps that hold the prosthesis to the body into a heavy-duty sports bra. The position of the harnessing straps are individualized for each woman so that the prosthesis can be positioned for optimal contact between the prosthetic sensor and the residual limb. The investigators foresee Brasthesis being available as an adaptable sports bra that comes with a goodie bag of spare parts that can be used to customize Brasthesis. The investigators plan to develop Brasthesis to be machine washable and relatively inexpensive so that Veterans can have more than one in a variety of colors.

DETAILED DESCRIPTION:
Current traditional prosthetic chest harnessing worn by women Veterans with limb loss) is less than optimal due to female anatomy. The investigators know from the sports and seat belt/airbag literature that breast tissue injuries can disrupt the blood flow to the breast resulting in swelling, significant blood loss, hematoma, fat necrosis, and oil cyst hematoma. Injury to the mammary ducts can affect the future or current flow of breast milk. More commonly, smaller superficial arteries along with veins become injured, leading to more localized injury and less serious bleeding and bruising. While there is no known research on whether a prosthetic harness can cause injury to breast tissue, the investigators know that frequent wearing of tight clothing can cause bruising, swelling, and thrombophlebitis. The investigators have designed a bra with incorporated prosthetic harness prototype for women Veterans with mid to short transhumeral, shoulder, or interscapulothoracic amputation(s) that the investigators have named Brasthesis (patent pending). The purpose of the proposed project is to use a case series design to prove the concept of Brasthesis prototype. The specific aims of this project are to: (1) Compare the satisfaction and function with and comfort of Brasthesis with the traditional harness and (2) Use pressure mapping to compare the interface pressure of Brasthesis with the traditional prosthesis. Five women with proximal upper limb loss will be fit with Brasthesis using a procedure similar to the one the investigators used for constructing the prototype. The inclusion criteria are: (1) unilateral mid to short trans-humeral, shoulder, or interscapular-thoracic unilateral amputation and (2) have an existing myoelectric or hybrid prosthetic limb that they used or rejected/abandoned. The additional resources required to train a participant with no prosthetic experience is judged beyond SPIRE resources/scope of this study. The exclusion criteria are: (1) open wounds in the upper torso or extremities and (2) body-powered prosthetic users due to the dynamic requirements of the harness. The investigators will pursue Using Brasthesis with body powered prosthetics in a subsequent study. Once the patient has provided written informed consent, two bras will be ordered. One bra the patient will wear. The second bra will be deconstructed and reconstructed for individualized suspensory harness strapping. At the time of Brasthesis fitting, baseline will be collected, demographic and clinical data and satisfaction, function, and comfort outcomes measures. After fitting, the participant will wear Brasthesis for four weeks. Participants will be contacted weekly to track wearing time in days per week and hours per day (Aim 1). The investigators will also employ a Jawbone Up 24 activity tracker as a quantitative proxy of prosthesis wear time. Pre to post ordinal change in wearing time, satisfaction, function, and comfort outcomes will be analyzed using quantitative descriptive analyses. At the end of the wearing period, PI Winkler will conduct semi-structured phone interviews with participants and the prosthetist. Interviews will be transcribed and analyzed using thematic analysis guided by descriptive phenomenology theory. The semi-structured interview will have three overall discussion points: (1) Describe the barriers encountered while fitting Brasthesis , (2) How did you manage strap placement based on the presence and length of the residual limb and the available skin surface area available for contact with the prosthetic sensor, and (3) How does Brasthesis compare with traditional prosthesis? Aim 2 will use pressure mapping technology to compare the residual limb and intact limb under arm pressure distribution data for Brasthesis and participants' traditional prostheses. The investigators will create color-coded 'heat maps' that directly link pressure values to the three-dimensional anatomy of each participant.

ELIGIBILITY:
Inclusion Criteria:

* mid to short transhumeral, shoulder, or interscapulothoracic unilateral amputation,
* have an existing myoelectric, hybrid, or cosmetic prosthetic limb that they use or have abandoned. The additional resources to train a participant with no prosthetic experience is beyond the scope of this study.

Exclusion Criteria:

* open wounds in the upper torso or extremities,
* body-powered prosthetic users are excluded due to the dynamic requirements of the harness. The investigators decided including women who did not have an existing prosthesis would exceed the time resources for a SPIRE funding mechanism.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Intervention includes wearing a sport bra. If a male with an upper limb amputation were to want to be fitted with a sports bra, he could be included in the study.
Enrollment: 5 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T Heckman, DO, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brasthesis
Started | 5
Participants Enrolled | 5
Completed | 4
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brasthesis
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
Socket Comfort Score [Mean (Standard Deviation); unit: units on a scale] — The Socket Comfort Score is a 1-item measure that rates comfort on a 11-point Likert-type scale with a range of 0-10. A higher score indicates more comfort.
  units on a scale | 4.8 (1.1)
Wear Time [Mean (Standard Deviation); unit: hours per week] | 32 (24.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Prosthetic Function and Satisfaction Using the Orthotic and Prosthetic Users Survey (OPUS)
Description: One of the OPUS self-report survey modules is the Upper Extremity Functional Status Survey which will be used to measure change:
  The Upper Extremity Functional Status Survey- when wearing a traditional and Brasthesis harness.
  1. The Upper Extremity Functional Status Survey has 28 items that are rated on a 5-point Likert type scale with a a possible range from 0 to 112 with a higher score representing a higher level of independent function.
Time Frame: Pre and post 4-week harness wearing time
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brasthesis
Number analyzed (Participants) | 4
Units on a scale | 73 (2.9)

2. Primary Outcome: Change in Comfort Measures With the Socket Comfort Score
Description: The change in comfort will be measured between the residual limb and socket and axilla of intact arm will be measured with the traditional harness (pre) ad Brasthesis (post).
  The Socket Comfort Score is a 1-item measure that rates comfort on a 11-point Likert-type scale with a range of 0-10. A higher score indicates more comfort.
Time Frame: Pre and post 4-week harness wearing time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brasthesis
Number analyzed (Participants) | 4
score on a scale | 4.75 (1.25)

3. Primary Outcome: Satisfaction With Devices
Description: The Satisfaction with Device Survey has 11 items that are rated on a 5-point Likert type scale with a a possible range from 11 to 55 with a higher score representing a better outcome, e.g., more satisfaction.
Time Frame: At post 4 week harness wearing time
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brasthesis
Number analyzed (Participants) | 4
units on a scale | 41.25 (5.8)

4. Secondary Outcome: Change in Range of Motion
Description: Change in range of motion of the residual limb will be measured using a goniometer.
  Normal values for shoulder flexion range from 0-180 Normal values for shoulder extension range from 0-60 Normal values for shoulder adduction range from 0-50 Normal values for shoulder abduction range from 0-180
Time Frame: Pre and post 4-week harness wearing time
Population: Two subjects were shoulder disarticulations and had no shoulder to measure shoulder range of motion from, so those two were excluded from analysis.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Brasthesis
Number analyzed (Participants) | 3
Degrees
  Change in ROM in shoulder flexion | 103 (56)
  Change in ROM in shoulder extension | 39 (18)
  Change in ROM in shoulder adduction | 0 (0)
  Change in ROM in shoulder abduction | 100 (53)

5. Secondary Outcome: Change in Pressure Using the Tekscan F-Socket Pressure Mapping System
Description: The change in pressure between the residual limb and socket and axilla of intact arm will be measured with the traditional harness (pre) ad Brasthesis (post). Data reported as mean max pressure mmHg
  Normal range of pressure readings are 0-250 mmHg
Time Frame: Pre and post 4-week harness wearing time
Population: Two subjects were not analysed. One withdrew and one had incomplete pressure mapping data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brasthesis
Number analyzed (Participants) | 3
mmHg | 92 (10)

6. Other Pre Specified Outcome: Activity Tracker
Description: The activity tracker measures prosthesis/harness wearing time and reports in 15 minute increments of time. Wearing time was summed to a calculation of hours per week across the 4 weeks of the study period. The range of hours per week is 0-168.
Time Frame: 4 week time frame from baseline to follow up
Measure: Mean (Standard Deviation); unit: Hours per week
Arm/Group | Brasthesis
Number analyzed (Participants) | 4
Hours per week | 43.75 (32.85)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Brasthesis
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT05179395/Prot_001.pdf
  • Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT05179395/SAP_002.pdf
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT05179395/ICF_000.pdf